CLINICAL TRIAL: NCT04226989
Title: A Study of CT-RD06 Cell Injection in Patients With Relapsed or Refractory CD19+ B-cell Hematological Malignancy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: He Huang (Other)
Collaborators: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, He Huang, Clinical Professor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-CT-RD06-03
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Acute Lymphoblastic Leukemia; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of CT-RD06 (Experimental): Dose escalation follows the standard 3+3 dose escalation design. A total of 3 dose levels are set for subjects.
  Interventions: Biological: CT-RD06

INTERVENTIONS:
Biological: CT-RD06 — CT-RD06 cell injection by intravenous infusion
  Other Names: CT-RD06 CAR-T cell injection

SUMMARY:
A study of CT-RD06 cell injection in patients with relapsed or refractory CD19+ B-cell hematological malignancy.

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study. This study is indicated for relapsed or refractory CD19+ B-cell hematological malignancy: B-ALL and B-NHL, the selections of dose levels and the number of subjects are based on clinical trials of similar foreign products. 2 groups of patients will be enrolled, 36 in each group. Primary objective is to explore the safety, main consideration is dose-related safety.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria only for B-ALL:

  1. Male or female aged 3-70 years;
  2. Histologically confirmed diagnosis of CD19+ B-ALL per the US National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Acute Lymphoblastic Leukemia (2016.v1);
  3. Relapsed or refractory CD19+ B-ALL (meeting one of the following conditions):

     1. CR not achieved after standardized chemotherapy;
     2. CR achieved following the first induction, but CR duration is ≤ 12 months;
     3. Ineffectively after first or multiple remedial treatments;
     4. 2 or more relapses;
  4. The number of primordial cells (lymphoblast and prolymphocyte) in bone marrow is﹥5% (by morphology), and/or﹥1% (by flow cytometry);
  5. Philadelphia-chromosome-negative (Ph-) patients; or Philadelphia-chromosome-positive (Ph+) patients who cannot tolerate TKI treatments or do not respond to 2 TKI treatments;
* Inclusion criteria only for B-NHL:

  1. Male or female aged 18-70 years;
  2. Histologically confirmed diagnosis of DLBCL (NOS), FL, DLBCL transformed from CLL/SLL, PMBCL, and HGBCL per the WHO Classification Criteria for Lymphoma (2016);
  3. Relapsed or refractory B-NHL (meeting one of the following conditions):

     1. No response or relapse after second-line or above chemotherapy regimens;
     2. Primary drug resistance;
     3. Relapse after auto-HSCT;
  4. At least one assessable tumor lesion per Lugano 2014 criteria;
* Common inclusion criteria for B-ALL and B-NHL:

  1. Total bilirubin ≤ 51 umol/L, ALT and AST ≤ 3 times of upper limit of normal, creatinine ≤ 176.8 umol/L;
  2. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥ 50%;
  3. No active infection in the lungs, blood oxygen saturation in indoor air is ≥ 92%;
  4. Estimated survival time ≥ 3 months;
  5. ECOG performance status 0 to 2;
  6. Patients or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

* Inclusion exclusion criteria only for B-ALL:

  1. Extramedullary lesions, except that CNSL (CNS-1) has been effectively controlled;
  2. Confirmed diagnosis of lymphoblastic crisis of chronic myeloid leukemia, Burkitt's leukemia/ lymphoma per WHO Classification Criteria;
  3. Hereditary syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome;
* Inclusion exclusion criteria only for B-NHL:

  1. Extranodal lesions in the brain (tumor cells in CSF, and/or MRI shows invasion of intracranial lymphoma);
  2. Extensive invasion of gastrointestinal lymphoma;
* Common exclusion criteria for B-ALL and B-NHL:

  1. History of hypersensitivity to any component of cell product;
  2. Prior treatment with any CAR T cell product or other genetically-modified T cell therapies;
  3. Prior treatment with radiotherapy, chemotherapy or mAb 1 week prior to apheresis;
  4. New York Heart Associate (NYHA) Class III/IV cardiac insufficiency (see Appendix 1);
  5. Myocardial infarction, cardioangioplasty or stenting, unstable angina pectoris, or other severe cardiac diseases within 12 months of enrollment;
  6. Severe primary or secondary hypertension of grade 3 or above (WHO Hypertension Guidelines, 1999);
  7. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
  8. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases;
  9. Severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
  10. Indwelling catheters in vivo (e.g. percutaneous nephrostomy, Foley catheter, bile duct catheter, or pleural/peritoneal/pericardial catheter). Ommaya storage, dedicated central venous access catheters such as Port-a-Cath or Hickman catheters are allowed;
  11. History of other primary cancer, except for the following conditions:

      1. Cured non-melanoma after resection, such as basal cell carcinoma of the skin;
      2. Cervical cancer in situ, localized prostate cancer, ductal cancer in situ with disease-free survival ≥ 2 years after adequate treatment;
  12. Autoimmune diseases requiring treatment, immunodeficiency or patients requiring immunosuppressive therapy;
  13. Prior immunizations with live vaccine 4 weeks prior to screening;
  14. History of alcoholism, drug abuse or mental illness;
  15. If HBsAg positive at screening, HBV DNA copy number detected by PCR in patients with active hepatitis B > 1000 (if HBV DNA copy number≤1000, routine antiviral therapy is required after enrollment), as well as CMV, hepatitis C, syphilis and HIV infection;
  16. Concurrent therapy with systemic steroids within 1 week prior to screening, except for the patients recently or currently receiving inhaled steroids;
  17. Patients who have participated in any other clinical studies within 2 weeks prior to screening;
  18. Female pregnant or lactating, male for female fertile but unable to take medically acceptable contraception measures;
  19. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-02-05 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CT-RD06 infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after CT-RD06 infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
B-cell acute lymphocytic leukemia(B-ALL), Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi ) at Month 6, 12, 18 and 24
B-ALL, Overall survival (OS) | Up to 2 years after CT-RD06 infusion
  From the first infusion of CT-RD06 to death or the last visit
B-ALL, Event-free survival (EFS) | Up to 2 years after CT-RD06 infusion
  From the first infusion of CT-RD06 to the occurrence of any event, including death, relapse or gene relapse, disease progression (any one occurs first), and the last visit
B cell non-hodgkin's lymphoma (B-NHL), Overall response rate (ORR) | At Week 4, 12, and Month 6, 12, 18, 24
  Assessment of ORR (ORR = CR + PR) per Lugano 2014 criteria
B-NHL, disease control rate (DCR) | At Week 12 and Month 6, 12, 18, 24
  Assessment of DCR (DCR=CR+PR+SD) per Lugano 2014 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Zhejiang Medical Colleage Zhejiang University, Hangzhou, Zhejiang, China